CLINICAL TRIAL: NCT01960335
Title: Whey Protein With and Without Exercise Training Enhances Total and Regional Body Composition, Insulin, Leptin, and Blood Pressure in Overweight and Obese Adults - The P+RISE Study
Brief Title: Whey Protein Intake With and Without Exercise on Visceral Fat: The P+RISE Study
Acronym: P+RISE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Skidmore College (Other)
Responsible Party: Principal Investigator, Paul Arciero, Professor, Health and Exercise Sciences Department, Director Human Nutrition and Metabolism Laboratory, Skidmore College
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: whey-1001-192
Record Dates: First submitted 2013-10-05; First posted 2013-10-10 (Estimated); Last update posted 2013-10-10 (Estimated); Status verified 2013-10

CONDITIONS: Obesity; Overweight
Keywords: whey protein intake; obesity; visceral fat; resistance exercise training; sprint interval training; endurance exercise training; yoga training; healthy eating; healthy lifestyle strategies; leptin; hunger
MeSH Terms: conditions — Obesity; Overweight | interventions — Whey Proteins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Whey Protein Only (Active Comparator): Ingestion of whey protein only (20 grams per serving) consumed 3X/day along with ad libitum diet for a total of 60 grams per day. One serving was consumed within 1 hour of waking in the morning; a second serving was consumed mid-afternoon; and a third serving was consumed within 2 hours of going to sleep at night.
  Interventions: Dietary Supplement: Whey Protein
- Whey Protein and Resistance Exericse (Experimental): Ingestion of whey protein (20 grams per serving) 3X/day: one serving within an hour of waking in morning; a second serving mid-afternoon or within 1 hour immediately following a resistance exercise bout on exercise days; and a third serving within 2 hours of going to bed at night.
  Interventions: Dietary Supplement: Whey Protein; Dietary Supplement: Whey Protein and Resistance Exericse
- Whey Protein and RISE exercise routine (Experimental): Ingestion of whey protein (20 gram serving) 3X/day: one serving within an hour of waking in the morning; a second serving mid-afternoon or within 1 hour immediately following the RISE exercise bout; and a third serving within 2 hours of going to bed at night.
  Interventions: Dietary Supplement: Whey Protein; Other: Whey Protein and RISE exercise routine

INTERVENTIONS:
Dietary Supplement: Whey Protein — Whey protein provided in 20 gram servings administered three times per day. once in the morning upon waking; a second serving in the mid-afternoon; and a third serving within 2 hours of going to sleep at night.
Dietary Supplement: Whey Protein and Resistance Exericse — Subjects will receive 20 grams of whey protein three times per day along with 4 days per week of resistance exercise training throughout the 16 week intervention.
  Arms: Whey Protein and Resistance Exericse
Other: Whey Protein and RISE exercise routine — Subjects will consume 20 grams of whey protein three times per day (total of 60 grams) and perform a combination of exercise involving functional resistance exercise (R); sprint intervals (I); stretching/pilates/yoga (S); and endurance exercise (E); RISE four days per week.
  Arms: Whey Protein and RISE exercise routine

SUMMARY:
Dietary manipulation is proving to be an effective lifestyle strategy to combat the obesity epidemic. Increased dietary protein is one effective strategy. For example, increased whey protein ingestion with and without exercise training is associated with enhanced weight loss, body composition and subjective hunger in overweight and obese individuals. Our findings suggest that the effects of whey protein ingestion occur independent of a calorie-restricted diet and to a greater extent in individuals following a combined exercise program of resistance exercise, sprint intervals, stretching/yoga/pilates, and aerobic exercise training compared to standard resistance training.

DETAILED DESCRIPTION:
This study was a 16 week whey protein and exercise training intervention in middle aged overweight/obese adults. Subjects were randomized into 3 groups: Whey protein only consumed as 20 grams per serving three times per day (total 60 grams per day) (WP); Whey protein and resistance exercise training (WP-RT); and Whey protein and combined exercise training (P+RISE). All outcomes, including the primary outcome of visceral fat was measured at baseline (week 0) and post-intervention (week 17) in all study subjects.

ELIGIBILITY:
Inclusion Criteria:

* healthy, overweight or obese, inactive

Exclusion Criteria:

* smoker, exercise-trained, recent weight loss, heavy caffeine-consumer

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 79 (Actual)
Dates: Start 2011-01; Primary Completion 2012-01 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
change in visceral fat | baseline and 17 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Paul J Arciero, Doctorate, Principal Investigator — Skidmore College
Locations (1):
- Health & Exercise Sciences Department, Human Nutrition and Metabolism Laboratory, Skidmore College, Saratoga Springs, New York, United States

REFERENCES:
- [Background] Baer DJ, Stote KS, Paul DR, Harris GK, Rumpler WV, Clevidence BA. Whey protein but not soy protein supplementation alters body weight and composition in free-living overweight and obese adults. J Nutr. 2011 Aug;141(8):1489-94. doi: 10.3945/jn.111.139840. Epub 2011 Jun 15. PMID 21677076